CLINICAL TRIAL: NCT02177097
Title: Extended Biochemical Analysis and Bacteriologic Diagnosis in Patients With Loose Joint Replacements, Chronic Pain and Infection.
Brief Title: Chronic Pain, Inflammation and Infection After Joint Replacement
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: N-20110022
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Infection and Inflammatory Reaction; Joint Prosthesis
Keywords: Pain; Infection; Inflammation; Prosthesis
MeSH Terms: conditions — Infections; Inflammation; Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 4 x 10 ml blood samples for each patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 40 patients (uTHA): Patients undergoing primary uncemented total hip arthroplasty surgery.
  Interventions: Biological: Blood samples
- 40 patients (hTHA): 40 patients undergoing primary hybrid total hip replacement surgery.
  Interventions: Biological: Blood samples
- 40 patients (TKA): 40 patients undergoing total knee replacement surgery.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — 4 x 10 ml blood samples.

SUMMARY:
Revision surgery after total hip or knee arthroplasty is an ongoing issue due to an increasing number of primary surgeries. Patients seek physicians due to pain. The cause is divided between loosening, infection or chronic pain. Some are operated on the suspicion of a chronic infection. However, postoperative microbiological testing does not always correlate with the suspicion and the operation may have been superfluous.

The objective is to employ a highly advanced diagnostic algorithm based on state of the art diagnostic techniques in order to improve the basis of preoperative diagnosis. Through this approach treatment can be given according to the causal problem.

DETAILED DESCRIPTION:
The aim of the project is to improve the preoperative diagnosis of infections and persistent pain in patients with prosthesis-related problems. Prosthesis infection is of chronic nature. Recent research has shown that one important explanation of this is the formation of encapsulated 'bacterial communities' on the surface of the prosthesis, where bacteria are well protected against antibiotic treatment. Surgery is therefore necessary for this patient group. But it is important to make diagnosis more accurate than it currently is today. In contrast, patients with persistent pain, but no indication of infection or prosthetic loosening, are best served by avoiding surgery, and instead receiving a treatment that is directed against the chronic pain condition. Based on the pain research carried out at Aalborg University, an understanding of chronic pain and treatment principles that would be beneficial for this patient group have been developed.

The investigators want to:

1. describe the postoperative course of specific serologic markers for primary and secondary total hip arthroplasty (THA) and total knee arthroplasty (TKA).
2. describe the bacteriologic diversity through revision of THA and TKA using cultivation techniques and molecular biological analysis comprehensive fluorescence in-situ hybridization (FISH), cloning and phylogeny, quantitative polymerase chain reaction (qPCR) and gene expression profiling.
3. describe pain and sensitization with new diagnostic technology in patients with stem loosening, suffering from infection and pain.
4. apply to a new diagnostic algorithm for the diagnosis of infection and pain following THA and TKA, which includes pain assessment, diagnostic X-ray, bone scintigraphy, PET scan, percutaneous biopsy, specific serologic parameters and molecular biological analysis.
5. describe the effect of the diagnostic algorithm, compared with a descriptive retrospective cohort of patients who have undergone revision of THA or TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary uncemented total hip-joint replacement surgery
* Patients undergoing primary hybrid total hip-joint replacement surgery
* Patients undergoing total knee-joint replacement surgery

Exclusion Criteria:

* Patients younger than 18 years old
* Unability to speak or read Danish
* Pregnancy or lactating
* Bilateral disease
* Cancer
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Examination of blood test parameters | 4 years
  The outcome measure is a composite.
  In order to predict the risk of developing a serious infection we want to:
  * develop serum concentration markers
  * describe bacteriological diversity
  * perform qualitative assessment of pain and sensitization

SECONDARY OUTCOMES:
Collect systematic data | 4 years
  The outcome measure is a composite. We want to collect systematic collect systematic data with a view to identify which specific blood parameters can best predict the risk that the patient develops a serious infection. Furthermore, we want to collect systematic data with a view to optimize the diagnostic algorithm.
Generate a knowledge base | 4 years
  The outcome measure is a composite. We want to generate a knowledge base for optimal antibiotic treatment, optimal pain management, optimal treatment of infection and pain caused by THA and TKA.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital
Locations (1):
- Northern Orthopaedic Division, Aalborg University Hospital, Aalborg, Denmark